CLINICAL TRIAL: NCT03173651
Title: The Efficiency of Different Oropharyngeal Airways as a Conduit for Fiberoptic Intubation. Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Sara Ahmed Abdallah, Assistant lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: N-40-2016
Record Dates: First submitted 2017-05-27; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Fiberoptic Tracheal Intubation

STUDY DESIGN:
Intervention Model Description: prospective randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group W (Experimental): This group was intubated by Fiberoptic bronchoscope assisted by Modified Williams airway as a conduit
  Interventions: Device: Modified Williams airway
- Group G (Experimental): This group was intubated by Fiberoptic bronchoscope assisted by Modified Guedle's airway as a conduit
  Interventions: Device: Modified Guedle's airway
- Group M (Experimental): This group was intubated by Fiberoptic bronchoscope assisted by LMA MADgic airway as a conduit
  Interventions: Device: LMA MADgic airway

INTERVENTIONS:
Device: Modified Williams airway — This airway used as a conduit for fiberoptic bronchoscopic tracheal intubation in Group W
  Other Names: Fikrey airway
  Arms: Group W
Device: Modified Guedle's airway — This airway used as a conduit for fiberoptic bronchoscopic tracheal intubation in Group G
  Arms: Group G
Device: LMA MADgic airway — This airway used as a conduit for fiberoptic bronchoscopic tracheal intubation in Group M
  Arms: Group M

SUMMARY:
60 Patients were randomly allocated into three equal groups, after induction of general anesthesia one of the three airways included in the study (Modified Williams, Modified Gudle's and LMA MADgic airway) was used as a conduit for endotracheal tube placement using fiberoptic bronchoscopy. Airway insertion time, ease of insertion, adaptation to oral cavity and intubation time was recorded.

DETAILED DESCRIPTION:
The study was conducted in Kasr Alainy hospital, faculty of medicine, Cairo University.

After approval of ethical committee and informed written consent from each patient, 60 patient aging above 18 years, ASA I-II , with Ganzouri airway score <4 and undergoing elective surgeries under general anesthesia were included in the study.

Patients were randomly allocated into three equal groups:

Group M (GM) (n=20 patients): patient was intubated using LMA MADgic airway. Group W (GW) (n=20 patients): patient was intubated using modified Williams airway.

Group G (GG) (n=20 patients): patient was intubated using modified Guedel's airway.

Randomization was performed by random computer allocation with numbered closed opaque envelopes.

The study was performed by expert anesthesiologist in FOB intubation. In the preparation room, all patients was cannulated with a 20 gauge venous cannula and 0.02mg/kg Midazolam was given. Patient transferred to the operating room and was monitored with non-invasive blood pressure, pulse oximetry and ECG. After preoxygenation using a facemask for 5 min, induction of anesthesia was done with 2mg/kg propofol, 1 μg/kg of fentanyl and 0.6 mg/kg of atracurium.

After loss of consciousness the selected airway according to group randomization was inserted into the mouth (size selection and technique of insertion according to manufacturer instruction). Time of insertion defined as the time, in seconds, from touching the patients' mouth with the airway until capnographic confirmation of ventilation by facemask. The ease of insertion was determined by number of attempts of airway insertion. Adaptation of the airway was determined by adequacy of ventilation, fitness to the oral cavity and appearance of successive ETco2 waves.

Manual positive-pressure ventilation was then started with 100% oxygen and 1-1.5% isoflurane through the facemask for 3 min until complete muscle relaxation was confirmed (when train-of-four count becomes zero).

Loaded FOB was inserted for intubation through the airway, laryngeal view grade was recorded (LVG) using Brimacomb and Berry scale; thereafter, the fiberscope was advanced into the trachea to a level just above the carina and the tracheal tube was railroaded over it.

Tracheal intubation could be facilitated by tube rotation, jaw thrust, neck extension or flexion and adjustment of the airway was allawed and was recorded. The intubation time was recorded ; that is, the time from cessation of manual ventilation using a facemask until restarting of ventilation through the tracheal tube.

The airway was removed except the LMA MADgic airway which was removed before ETT insertion. The ease of airway removal was evaluated by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical state I-II Ganzouri airway score less than 4

Exclusion Criteria:

* ASA physical state III-IV. Patients with Ganzouri airway score more than 4. Patients with risk of aspiration of gastric content. Any anatomical abnormalities or iatrogenic injuries that invalidate Ganzouri airway score.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time of intubation | within 15 minutes from induction of general anesthesia
  The time from cessation of manual ventilation using a facemask until restarting of ventilation through the tracheal tube

SECONDARY OUTCOMES:
Time of insertion | within 15 minutes from induction of general anesthesia
  Time from touching the patients' mouth with the airway until capnographic confirmation of ventilation by facemask
Laryngeal View Grade | within 15 minutes from induction of general anesthesia
  Degree of vocal cord visualization by fiberoptic bronchoscope

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ahmed Abdallah, Master, Principal Investigator — Kasr El Aini Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dina N. Abbas, Ekramey M. Abdghaffar. Comparison of the air-Q intubating laryngeal airway versus the modified Williams intubating airway as aids for training in fiberoptic tracheal intubation. Ain-Shams Journal of Anesthesiology 2013, 6:134-139.